CLINICAL TRIAL: NCT05063123
Title: A Phase II Multicenter Study to Assess the Feasibility and Efficacy of the Addition of an Interphase Cycle With Flotetuzumab Prior to Start Conditioning for an Allogeneic HCT in AML With MRD After 2 Cycles of Intensive Chemotherapy
Brief Title: Study to Assess an Interphase Cycle With Flotetuzumab.
Acronym: HOVON162AML
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawal of MacroGenics (pharmaceutical company)
Sponsor: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HO162; 2021-001041-12 (EudraCT Number)
Record Dates: First submitted 2021-09-13; First posted 2021-09-30 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-09

CONDITIONS: AML
Keywords: MRD positive; APL excluded

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm - Flotetuzumab (Other): 1 - 3 cycles of Flotetuzumab. Flotetuzumab will be administered intravenously via continuous (pump) administration. At least for the first 7 days of cycle 1, the drug will be administered in an inpatient hospital setting, but afterwards may be administered in an outpatient setting using an ambulatory pump configuration. Flotetuzumab will be dosed using multi-step increments in dosing over the first week as follows: 30, 60, 100, 200, 300, and 400 ng/kg/day each for 24 hours. On day 7, the dose will be increased to 500 ng/kg/day and administered as a continuous infusion for the remainder of cycle 1. After 1 cycle of flotetuzumab patients will proceed with alloHCT. However if there is a delay in access to transplantation, patients are allowed to receive up to 2 additional cycles flotetuzumab provided all non-hematologic toxicities have resolved to Grade <2.
  Interventions: Drug: Flotetuzumab

INTERVENTIONS:
Drug: Flotetuzumab — Flotetuzumab will be given after at least 2 intensive chemotherapy cycles and before the start of the conditioning regimen prior to allo-HCT.

SUMMARY:
Patients who have measurable residual disease (MRDpos, defined as MRD > 0.1% by flowcytometry or detectable mutant Nucleophosmin 1 (NPM1) by quantitative polymerase chain reaction (qPCR) after two cycles of intensive chemotherapy) prior to start conditioning for an allogeneic Hematopoietic Cell Transplantation (HCT) have a very high risk of relapse after transplantation. Important questions in the field are whether patients with MRD after intensive chemotherapy can be converted to MRD negativity (i.e. undetectable MRD, MRDneg) and whether this conversion impacts on the relapse rate after transplantation. This trial aims to develop effective "interphase" treatment for patients in morphological complete remission (CR) with MRD after at least 2 cycles of intensive chemotherapy and prior to start conditioning for an allogeneic HCT. Flotetuzumab, a bispecific antibody-based molecule against CD3 and CD123 in a dual-affinity re-targeting antibody (DART®) format is a new treatment modality based on immunomodulation. The rationale to use flotetuzumab in this study is: 1) its antileukemic activity reported in R/R AML; 2) its limited extra-medullary (i.e. tissue) toxicity; and 3) its short halflife.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Diagnosis of ELN AML other than acute promyelocytic leukemia (APL) with t(15;17)(q22;q12) or variants of these according to the 2016 WHO classification.
* In first CR/CRi/CRh after at at least 2 cycles of intensive chemotherapy with MRD by l MFC-based MRD assay or qPCR mutant NPM1 assessed by central lab. Three cycles of intensive treatment is allowed if 2 cycles of treatment were needed to reach morphological remission.
* Should be off any active systemic therapy for AML for at least 14 days or 5 half-lives (whichever is longer) prior to study registration
* All Grade 2-4 non-hematologic toxicities should have resolved.
* Planned to undergo myeloablative or reduced intensity conditioning prior to alloHCT with a likely source for donor cells identified.
* Eastern Cooperative Oncology Group (ECOG)/ WHO performance status 0-2.
* Adequate hepatic and renal function

  * Both alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels (less or equal then) 2.5 times the institutional upper limit of normal (ULN).
  * Total bilirubin level (less or equal then) 1.5 times the ULN (unless the patient has a history of Gilbert's Syndrome, in which case, total bilirubin must be (less or equal then) 2.5 times the ULN).
  * Serum creatinine level (less or equal then) 1.5 times the ULN or a calculated or measured creatinine clearance of ≥ 50 mL/min.
* Adequate organ reserve including cardiovascular, pulmonary, renal, and hepatic functioning sufficient, in the judgment of the Investigator, to undergo therapy.

  - If there is a history or signs of heart failure, an echocardiography or MUGA should be obtained, with the estimated left ventricular ejection fraction required to be ≥45%.
* Women of childbearing potential must test negative for pregnancy at enrollment.
* Sexually active women of child-bearing potential must be willing to use a highly effective method of birth control from the time of consent through 12 weeks after flotetuzumab administration. A highly effective method is defined as those which result in a low failure rate (i.e., less than 1% per year) such as implants, injectables, combined oral contraceptives, intra-uterine devices (IUDs) or vasectomized partner.
* Male patients with partners of childbearing potential must be either vasectomized or agree to use a condom in addition to having their partners use another method of contraception resulting in a highly effective method of birth control defined as those which result in a low failure rate (i.e., less than 1% per year) such as implants, injectables, combined oral contraceptives, or IUDs. Patients should not have sexual intercourse with females who are either pregnant or lactating without double barrier contraception. Contraception should be employed from the time of consent through 12 weeks after flotetuzumab administration.
* Patient is able and willing to adhere to the study visit schedule and other protocol requirements.
* Patient is capable of giving informed consent.
* Written informed consent.

Exclusion Criteria:

* Prior history of allogeneic HCT.
* Prior treatment with an anti-CD123-directed agent.
* Favorable risk AML other than AML with NPM1 mutation (according to 2017 ELN)
* Myeloid blast crisis of chronic myeloid leukemia (CML).
* Concomitant illness associated with an estimated survival of <1 year.
* Any active untreated autoimmune disorders (with the exception of vitiligo, resolved childhood atopic dermatitis, prior Grave's disease now euthyroid clinically and with stable supplementation).
* Second primary malignancy that requires active therapy. Adjuvant hormonal therapy is allowed. Patients with the following history/concurrent conditions are allowed:

  * Basal or squamous cell carcinoma of the skin
  * Carcinoma in situ of the cervix
  * Carcinoma in situ of the breast
  * Incidental histologic finding of prostate cancer
* Active systemic fungal, bacterial, viral, or other infection, unless disease is under treatment with anti-microbials, and/or controlled or stable (e.g. if specific, effective therapy is not available/feasible or desired [e.g. chronic viral hepatitis, HIV]). Patient needs to be clinically stable as defined as being afebrile and hemodynamically stable for 24 hours.
* Requirement, at the time of study entry, for concurrent steroids >10 mg/day of oral prednisone or the equivalent, except steroid inhaler, nasal spray or ophthalmic solution.
* Use of immunosuppressant medications (other than steroids as noted) in the 2 weeks prior to study drug administration.
* Use of granulocyte colony stimulating or granulocyte-macrophage colony stimulating factor in the 2 weeks prior to study drug administration.
* Known central nervous system (CNS) leukemia. Patients with suspected CNS leukemia must be evaluated by lumbar puncture and be free of CNS disease prior to study entry. Previously treated CNS leukemia is allowed provided adequate treatment has been provided and the patient is free of CNS disease.
* Known hypersensitivity to murine, yeast, or recombinant proteins; polysorbate 80; recombinant human serum albumin; benzyl alcohol; or any excipient contained in the flotetuzumab drug formulation.
* Dementia or altered mental status that would preclude sufficient understanding to provide informed consent.
* Pregnant or lactating female patient.
* Current participation in another clinical trial.
* Any psychological, familial, sociological and geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of CR/CRi without MRD defined as MRD < 0.1% by flowcytometry or undetectable mutant NPM1 by qPCR after 1 cycle of flotetuzumab | 1 year after inclusion last patient
  The primary objective of this study is to assess the rate of MRDneg remission after treatment with one cycle of flotetuzumab.
  The rate of MRDneg remission after one treatment cycle will be tabulated and exact 95% confidence intervals will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: M. Jongen-Lavrencic, PhD, Principal Investigator — Erasmus Medical Center
Locations (4):
- Netherlands (4):
  - NL-Amsterdam-VUMC, Amsterdam
  - NL-Groningen-UMCG, Groningen
  - NL-Maastricht-MUMC, Maastricht
  - NL-Rotterdam-ErasmusMC, Rotterdam

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with Fred Hutchinson / University of Washington Cancer Consortium
Supporting Information: Study Protocol, SAP

REFERENCES:
- See also: HOVON website — http://www.hovon.nl